CLINICAL TRIAL: NCT05538377
Title: Effect of Focal Vibration on Bone Quality Within a Multicomponent Exercise Program for Older Women With Osteoporosis a Single-blind Clinical Trial
Brief Title: Effect of Focal Vibration Within a Multicomponent Exercise Program for Older Women With Osteoporosis a Single-blind Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jacobo Rodríguez Sanz, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFC22OST
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Osteoporosis; Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focal Vibration (Experimental)
  Interventions: Other: Focal Vibration
- Control Group (Active Comparator)
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Focal Vibration — This group will receive a multicomponent exercise program based on specific literature for effective training. In addition, this group will perform the strength and endurance exercises with focal vibration on the vastus internus, externus and biceps femoris. There will be 2 sessions per week, with a duration of 60 minutes per session and a treatment duration of 6 months.
  Arms: Focal Vibration
Other: Control Group — This group will receive the same multicomponent exercise program than the other group based on specific literature for effective training. There will be 2 sessions per week, with a duration of 60 minutes per session and a treatment duration of 6 months.
  Arms: Control Group

SUMMARY:
The high annual incidence of osteporosis and its high prevalence , means that more and more resources are being devoted to its diagnosis, prevention and treatment in primary care. This pathology is defined as a skeletal disorder characterized by an alteration in bone strength, mainly reflecting a poor integration of bone density and quality.

The reduction of the mass and the alteration of the microstructure of osteoporotic bone lead to an increase in its fragility and an increase in the risk of suffering bone fractures. If we add to this the alterations in balance observed in older people, the possibility of fracture and increased fragility increases. It is estimated that every 3 seconds there is an osteoporotic fracture and it is considered that every year 8.9 million fractures of this type occur worldwide. Fragility fractures are estimated to be associated with significant morbidity and mortality. In the case of hip fracture as a consequence of osteoporosis, only 30-45% of surviving cases recover pre-fracture functional status and 32-80% suffer some form of significant dysfunction, thus representing a high economic and social cost.

Associated with osteoporosis, numerous studies have also observed a decrease in strength and/or muscle mass (sarcopenia), thus increasing the fragility and deterioration of the patient suffering from osteoporosis. Tokeshi et al. observed that patients with osteoporotic fractures had less muscle mass compared to patients without osteoporosis. Hoo Lee and Sik Gong describe that lower extremity muscle mass and loss of grip are closely related to the occurrence of an osteoporotic vertebral fracture and numerous investigations show the relationship between grip strength and osteoporotic fractures in the elderly.

For the diagnosis of osteoporosis, double beam X-ray densitometry (DEXA) is used and osteoporosis is considered to be present when the osteoporosis values are below 2.5 standard deviations (SD) of the peak bone mass, the maximum value reached in young women.

At the therapeutic level, pharmacology is the treatment recommended in clinical practice guidelines. However, due to poor adherence and adverse effects, the recommendation of physical activity programs is becoming more and more popular to increase mineral density and bone quality, either as adjuvant treatments or as the treatment of choice.

Various research and clinical guidelines recommend the use of therapeutic exercise as part of the treatment of osteoporosis. The National Osteoporosis Foundation of the United States concludes that the practice of exercise improves, among other benefits, the quality of bone mass. Likewise, different systematic reviews have shown that multicomponent training in older people is effective in preventing or maintaining bone mass, especially when such exercises are performed with high load or high impact or when performed by postmenopausal women.

Along these lines, the American College of Sports Medicine and recent research demonstrates how strength work at moderate to high load intensity can not only stimulate bone metabolism, but also improve the quality of life of those who practice it.

But in spite of the bone benefit observed with high loads for bone tissue, not all elderly people can do it, either because of the fragility that many of them present, or because of the mechanical stress that this type of exercise produces in their joints. For this reason, one of the possible alternatives that we have found for some decades is training through the use of global vibration (GV) or body vibration through the use of vibrating platforms. This type of vibration generally starts in the extremities and the limbs themselves are used as a sounding board for the vibrational stimulus to the rest of the body. This type of equipment has allowed a less demanding training from the articular point of view in a less demanding approach to other exercise programs in patients and has shown significant improvements in bone formation rate, bone mineral density (BMD), trabecular structural and cortical thickness in osteporotic bone tissue.

But despite the wide use of vibrating platforms for training in elderly people, it is not free of contraindications such as patients with recent fracture, deep vein thrombosis, osteosynthesis of lower limbs, hip prosthesis, aortic aneurysm or diabetic foot injury, for this reason have emerged focal vibration devices (VF). This tool allows the application of the vibratory stimulus in a specific and repeated way in a part of the body; as well as the control of the amplitude that reaches a certain tissue avoiding the disadvantages of the vibratory platforms in which the region and the tissue to be treated cannot be selected.

DETAILED DESCRIPTION:
The high annual incidence of osteporosis (1% in women aged 65 years, 2% in women aged 75 years and 3% in women over 85 years) and its high prevalence (30% in postmenopausal women), means that more and more resources are being devoted to its diagnosis, prevention and treatment in primary care. According to the World Health Organization (WHO), this pathology is defined as a skeletal disorder characterized by an alteration in bone strength, mainly reflecting a poor integration of bone density and quality. Primary (or also known as idiopathic) osteoporosis can affect both sexes, but postmenopausal and older women are more vulnerable.

The reduction of the mass and the alteration of the microstructure of osteoporotic bone lead to an increase in its fragility and an increase in the risk of suffering bone fractures. If we add to this the alterations in balance observed in older people, the possibility of fracture and increased fragility increases. It is estimated that every 3 seconds there is an osteoporotic fracture and it is considered that every year 8.9 million fractures of this type occur worldwide. Fragility fractures are estimated to be associated with significant morbidity and mortality. In the case of hip fracture as a consequence of osteoporosis, only 30-45% of surviving cases recover pre-fracture functional status and 32-80% suffer some form of significant dysfunction, thus representing a high economic and social cost.

Associated with osteoporosis, numerous studies have also observed a decrease in strength and/or muscle mass (sarcopenia), thus increasing the fragility and deterioration of the patient suffering from osteoporosis. Tokeshi et al. observed that patients with osteoporotic fractures had less muscle mass compared to patients without osteoporosis. Hoo Lee and Sik Gong describe that lower extremity muscle mass and loss of grip are closely related to the occurrence of an osteoporotic vertebral fracture and numerous investigations show the relationship between grip strength and osteoporotic fractures in the elderly.

For the diagnosis of osteoporosis, double beam X-ray densitometry (DEXA) is used and osteoporosis is considered to be present when the osteoporosis values are below 2.5 standard deviations (SD) of the peak bone mass, the maximum value reached in young women.

At the therapeutic level, pharmacology is the treatment recommended in clinical practice guidelines. However, due to poor adherence and adverse effects, the recommendation of physical activity programs is becoming more and more popular to increase mineral density and bone quality, either as adjuvant treatments or as the treatment of choice.

Various research and clinical guidelines recommend the use of therapeutic exercise as part of the treatment of osteoporosis. The National Osteoporosis Foundation of the United States concludes that the practice of exercise improves, among other benefits, the quality of bone mass. Likewise, different systematic reviews have shown that multicomponent training in older people is effective in preventing or maintaining bone mass, especially when such exercises are performed with high load or high impact or when performed by postmenopausal women.

Along these lines, the American College of Sports Medicine and recent research demonstrates how strength work at moderate to high load intensity can not only stimulate bone metabolism, but also improve the quality of life of those who practice it.

But in spite of the bone benefit observed with high loads for bone tissue, not all elderly people can do it, either because of the fragility that many of them present, or because of the mechanical stress that this type of exercise produces in their joints. For this reason, one of the possible alternatives that we have found for some decades is training through the use of global vibration (GV) or body vibration through the use of vibrating platforms. This type of vibration generally starts in the extremities and the limbs themselves are used as a sounding board for the vibrational stimulus to the rest of the body. This type of equipment has allowed a less demanding training from the articular point of view in a less demanding approach to other exercise programs in patients and has shown significant improvements in bone formation rate, bone mineral density (BMD), trabecular structural and cortical thickness in osteporotic bone tissue.

But despite the wide use of vibrating platforms for training in elderly people, it is not free of contraindications such as patients with recent fracture, deep vein thrombosis, osteosynthesis of lower limbs, hip prosthesis, aortic aneurysm or diabetic foot injury, for this reason have emerged focal vibration devices (VF). This tool allows the application of the vibratory stimulus in a specific and repeated way in a part of the body; as well as the control of the amplitude that reaches a certain tissue avoiding the disadvantages of the vibratory platforms in which the region and the tissue to be treated cannot be selected.

ELIGIBILITY:
Inclusion Criteria:

* A woman between 60 and 75 years of age with a medical diagnosis of osteoporosis by means of a femur or lumbar densitometry of less than 2.5 standard deviations (SD) of peak bone mass.
* No history of previous fracture in the last 10 years.

Exclusion Criteria:

* Secondary osteoporosis.
* Having suffered a bone fracture in the last year.
* Having had juvenile osteoporosis during adolescence or young adulthood.
* Uncontrolled arterial hypertension.
* Uncontrolled orthostatic hypotension.
* Severe acute respiratory failure.
* Diabetes mellitus with acute decompensation or uncontrolled hypoglycemia.
* Endocrine, hematological and other associated rheumatic diseases.
* Mental health problems (schizophrenia, dementia, depression, etc.) or not being in full mental capacity.
* Patients with pharmacological treatments of glucocorticoids, anticoagulants and/or diuretics.
* Patients with coagulation problems or previous cardiac pathology.
* People with a body mass index (BMI) equal to or higher than 30.
* Subjects who present a systemic disease or any other pathology in which therapeutic exercise could be contraindicated.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with osteoporosis
Enrollment: 34 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in bone mineral density (mg/cm3) | Baseline; 6 months follow-up; 9 month follow-up; 1 year follow-up; 15 months follow-up
  Bone mineral density will be analyzed by radiological densitometry using quantitative ultrasound. This technique is completely harmless to the patient and has been shown in numerous investigations to predict the risk of osteoporotic fractures.

SECONDARY OUTCOMES:
Senior Fitness test (questionnaire) | Baseline; 6 months follow-up; 9 month follow-up; 1 year follow-up; 15 months follow-up
  Consists of a battery of tests specifically designed for the elderly population to assess their functional condition to perform normal activities of daily living safely, independently and without excessive fatigue.
30-m walk test (seconds) | Baseline; 6 months follow-up; 9 month follow-up; 1 year follow-up; 15 months follow-up
  The maximum walking speed will be measured by the 30-m walk test, which measures the time spent walking 30 m as fast as possible without running.
Chair stand test (attempts) | Baseline; 6 months follow-up; 9 month follow-up; 1 year follow-up; 15 months follow-up
  Lower extremity strength will be measured with the chair stand test, which will measure the number of times the person can stand up and sit down in a chair in 30 s.
Arm curl test (attempts) | Baseline; 6 months follow-up; 9 month follow-up; 1 year follow-up; 15 months follow-up
  Upper extremity strength was measured with the arm curl test, in which the elderly had to lift a 4 kg (men) or 2.5 kg (women) dumbbell to the maximum number of repetitions in 30 s.
Maximum isometric strength (Newtons) | Baseline; 6 months follow-up; 9 month follow-up; 1 year follow-up; 15 months follow-up
  Maximum isometric strength of the lower and upper extremity will be assessed using a manual dynamometer.
Handgrip (Newtons) | Baseline; 6 months follow-up; 9 month follow-up; 1 year follow-up; 15 months follow-up
  The participant must squeeze the dynamometer as hard as possible and the force applied will be recorded.
Balance Surface (mm2) | Baseline; 6 months follow-up; 9 month follow-up; 1 year follow-up; 15 months follow-up
  The surface comprises 95% of all the measured points of the center of pressures. It is measured in square millimeters. A larger surface area of the ellipse implies a lower capacity to maintain equilibrium at the center of pressure.
Balance length (mm) | Baseline; 6 months follow-up; 9 month follow-up; 1 year follow-up; 15 months follow-up
  It is measured in millimeters, and assesses the accuracy of the fine postural system in maintaining balance. A longer stabilogram length indicates a greater involvement of the fine control system in rebalancing.
Frail Scale | Baseline; 6 months follow-up; 9 month follow-up; 1 year follow-up; 15 months follow-up
  Is a 5-item questionnaire that measures fatigue (in the last 4 weeks), endurance (being able to climb 10 steps without resting), ambulation (having some difficulty walking hundreds of meters), illness and body weight loss during the last year.
SF-36 (questionnaire 0-100) | Baseline; 6 months follow-up; 9 month follow-up; 1 year follow-up; 15 months follow-up
  The items are coded, aggregated and transformed into a scale ranging from 0 (the worst health status for that dimension) to 100 (the best health status).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain